CLINICAL TRIAL: NCT00573508
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 4, Multi-center Study of VESIcare® (Solifenacin Succinate) in Overactive Bladder (OAB) Subjects to Evaluate Symptom Bother and Health Related Quality of Life VIBRANT: VESIcare® Investigation of BotheR And Quality of Life iN subjecTs With OAB
Brief Title: Study of VESIcare® In Overactive Bladder (OAB) Subjects to Evaluate Symptom Bother and Health Related Quality of Life
Acronym: VIBRANT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr. Manager Clinical Trials Registry, Astellas Pharma US, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 905-UC-010
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Active Comparator): Matching placebo tablet taken once daily
  Interventions: Drug: Placebo
- Solifenacin Succinate (Experimental): 5mg or 10mg tablet taken once daily
  Interventions: Drug: Solifenacin Succinate

INTERVENTIONS:
Drug: Placebo — Oral Administration
  Arms: Placebo
Drug: Solifenacin Succinate — Oral Administration
  Other Names: VESIcare®; YM905
  Arms: Solifenacin Succinate

SUMMARY:
Evaluate the effect of VESIcare® on symptom bother for subjects with OAB

DETAILED DESCRIPTION:
Phase 4, multi-center, randomized, double-blind, placebo-controlled, parallel group study. All subjects that meet the baseline criteria will be randomized in a 1:1 ratio into VESIcare® (solifenacin succinate) or placebo group.

The study duration consists of a screening period which includes a minimum of a 14 day treatment free wash-out period. Subjects meeting the baseline criteria will have a 12 week treatment period. Maximum total study duration is 15 weeks: 2 3 week screening / washout period; 12 week double-blind treatment.

Primary efficacy will be based on OAB-q symptom bother score.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female subject ≥ 18 years of age and able to use the toilet without difficulty
* History of OAB symptoms for ≥ 3 months
* An average of ≥ 8 micturitions per 24 hours and ≥ 1 urgency episode (with or without incontinence) per 24 hours as documented in a 3-day micturition diary
* Subjects are bothered by symptoms as reflected by PPBC ≥3

Exclusion Criteria:

* Evidence of chronic urologic inflammation such as interstitial cystitis and bladder stones; uncontrolled narrow angle glaucoma; urinary or gastric retention
* Recurrent urinary tract infection (UTI) of > 3 episodes within the last 3 months or evidence of a urinary tract infection at Baseline Visit (Visit 2)
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the investigator
* History of renal or hepatic impairment(2 x Upper Limit of Normal(ULN) values in parameters and considered clinically significant by the investigator
* History of diagnosed gastrointestinal obstruction disease
* Subject has a known diagnosis or history of carcinoma (including prostate cancer) except non metastatic basal or squamous cell carcinoma of the skin that has been successfully treated or previous pelvis radiation within the past five years
* Known or suspected hypersensitivity to solifenacin succinate, any components, or other anticholinergics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (56):
- United States (56):
  - Montgomery, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Buena Park, California
  - Carmichael, California
  - Fresno, California
  - Sacramento, California
  - San Bernardino, California
  - San Diego, California
  - Aurora, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - Waterbury, Connecticut
  - Clearwater, Florida
  - Plantation, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Roswell, Georgia
  - Idaho Falls, Idaho
  - Melrose Park, Illinois
  - Jeffersonville, Indiana
  - Shreveport, Louisiana
  - Watertown, Massachusetts
  - Billings, Montana
  - Omaha, Nebraska
  - Englewood, New Jersey
  - Lawrenceville, New Jersey
  - Endwell, New York
  - Garden City, New York
  - Kingston, New York
  - New York, New York
  - Orchard Park, New York
  - Poughkeepsie, New York
  - Concord, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Lyndhurst, Ohio
  - Edmond, Oklahoma
  - Central Point, Oregon
  - Philadelphia, Pennsylvania
  - Uniontown, Pennsylvania
  - West Reading, Pennsylvania
  - Greer, South Carolina
  - Simpsonville, South Carolina
  - Arlington, Texas
  - Austin, Texas
  - Bedford, Texas
  - Corpus Christi, Texas
  - Houston, Texas
  - Mount Lake, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin

REFERENCES:
- [Result] Vardy MD, Mitcheson HD, Samuels TA, Wegenke JD, Forero-Schwanhaeuser S, Marshall TS, He W. Effects of solifenacin on overactive bladder symptoms, symptom bother and other patient-reported outcomes: results from VIBRANT - a double-blind, placebo-controlled trial. Int J Clin Pract. 2009 Dec;63(12):1702-14. doi: 10.1111/j.1742-1241.2009.02209.x. PMID 19930331
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Crosby RD, Mathias SD, Marshall TS. Relationships between symptoms, symptom bother, and health-related quality of life in patients with overactive bladder taking solifenacin or placebo in the VIBRANT study. Int J Clin Pract. 2011 Feb;65(2):211-8. doi: 10.1111/j.1742-1241.2010.02532.x. PMID 21235700
- See also: Link to Prescribing Information — http://www.astellas.us/docs/vesicare.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Solifenacin Succinate
Started | 382 | 386
Full Analysis Set (FAS) | 374 (Patients who took >= 1 dose of double-blind study drug, had a baseline OAB-q & >= 1 subsequent visit) | 377 (Patients who took >= 1 dose of double-blind study drug, had a baseline OAB-q & >= 1 subsequent visit)
Completed | 318 | 345
Not Completed | 64 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Solifenacin Succinate | Total
Number analyzed (Participants) | 382 | 386 | 768
Age Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.36) | 59.4 (13.44) | 59.4 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 321 | 311 | 632
  Male | 61 | 75 | 136
Race/Ethnicity, Customized [Number; unit: participants]
  White | 333 | 347 | 680
  Black or African American | 30 | 24 | 54
  Asian | 9 | 7 | 16
  American Indian or Alaska Native | 3 | 3 | 6
  Native Hawaiian-Other Pacific Islander | 0 | 1 | 1
  Other | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment in Overactive Bladder Questionnairre (OAB-q) Symptom Bother Score
Description: The OAB-q is used to assess how much a patient is bothered by OAB symptoms & the impact of these symptoms on the patient's Health Related Quality of Life(HRQL). It is a patient administered tool comprised of 33 items, where the first 8 define symptom bother with raw score being converted to a scale of 0 to 100.
  Higher score values are indicative of greater symptom severity or bother, and a lower score in change from baseline indicates improvement.
  End of Treatment results include patients who had early discontinuation from the study.
  Change is calculated as End of Treatment - Baseline.
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set(FAS): all randomized patients who took at least 1 dose of double-blind study medication and had an assessment in OAB-q at both baseline and at least 1 post-baseline visit.
  The number of participants per arm is consistent for all categories / rows of the data table.
Measure: Mean (Standard Deviation); unit: OAB-q Score
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
OAB-q Score
  Baseline | 57.9 (18.18) | 58.2 (18.75)
  End of Treatment | 37.5 (22.54) | 28.3 (20.36)
  Change at End of Treatment | -20.4 (21.72) | -29.9 (22.64)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Statistical Analysis applies to 'Change at End of Treatment'; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Square Mean Difference = 9.4, 95% CI [6.6 to 12.2]

2. Secondary Outcome: Change From Baseline to Each Visit in Symptom Bother Utilizing the OAB-q Score
Description: The OAB-q is used to assess how much a patient is bothered by OAB symptoms and the impact of these symptoms on the patient's HRQL. It is a validated patient administered tool comprised of 33 items, where the first 8 items define symptom bother with raw score being converted to a scale of 0 to 100.
  Higher score values are indicative of greater symptom severity or bother, and a lower score in change from baseline indicates improvement.
  Change is calculated as Actual Data for each timepoint - Baseline.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: Population is full analysis set(FAS): all randomized patients who took at least 1 dose of double-blind study medication and had an assessment in OAB-q at both baseline and at least 1 post-baseline visit.
  The number of participants analyzed per arm represents FAS. The numbers of participants for each visit are noted in the category titles.
Measure: Mean (Standard Deviation); unit: OAB-q Score
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
OAB-q Score
  Baseline ( N= 374 ; 377) | 57.9 (18.18) | 58.2 (18.75)
  Week 4 (N=371; 370) | 41.6 (21.04) | 35.5 (20.77)
  Change at Week 4 (N=371; 370) | -16.4 (19.33) | -22.6 (20.55)
  Week 8 (N=342; 356) | 37.0 (21.86) | 29.8 (20.23)
  Change at Week 8 (N=342; 356) | -21.0 (20.64) | -28.9 (22.11)
  Week 12 (N=318; 339) | 36.0 (21.91) | 27.6 (20.32)
  Change at Week 12 (N=318; 339) | -21.7 (21.52) | -30.9 (22.29)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Statistical Analysis applies to 'Change at Week 4', 'Change at Week 8' and 'Change at Week 12'; Test type: Superiority or Other; p < .0001, ANCOVA

3. Secondary Outcome: Change From Baseline to Each Visit in OAB-q Health Related Quality of Life (HRQL) Total Score
Description: The OAB-q is used to assess how much a patient is bothered by OAB symptoms and the impact of these symptoms on the patient's HRQL. It is a validated patient administered tool comprised of 33 items, where items 9 - 33 define HRQL with raw score being converted to a scale of 0 to 100.
  Higher score values are indicative of better HRQL, and a positive score in change from baseline indicates improvement.
  Change is calculated as Actual Data for each time point - Baseline.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: OAB-q HRQL Total Score
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
OAB-q HRQL Total Score
  Baseline (N= 374 ; 377) | 57.8 (21.34) | 56.4 (22.10)
  Week 4 (N=371; 370) | 71.4 (21.42) | 76.0 (20.81)
  Change at Week 4(N=371; 370) | 13.5 (17.92) | 19.3 (19.43)
  Week 8 (N=342; 356) | 75.2 (21.06) | 80.5 (19.94)
  Change at Week 8 (N=342; 356) | 17.3 (19.00) | 24.4 (21.35)
  Week 12 (N=318; 339) | 76.7 (20.53) | 82.2 (19.64)
  Change at Week 12(N=318; 339) | 18.0 (19.39) | 25.8 (22.30)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Statistical Analysis applies to 'Change at Week 12'; Test type: Superiority or Other; p < .0001, ANCOVA — P-Value represents change from Baseline to Week 12

4. Secondary Outcome: Number of Participants With Change From Baseline in the Global Assessment Score of the Patient Perception of Bladder Condition (PPBC)
Description: The PPBC is a validated, global assessment tool using a 6-point Likert scale which requires patients to assess their bladder condition by selecting one of the following responses: 1=Does not cause me any problem at all; 2=Cause me some very minor problems; 3=Causes me some minor problems; 4=Causes me (some) moderate problems; 5=Causes me severe problems; 6=Causes me many severe problems
  Improvement is defined by any reduction in PPBC score.
  End of Treatment results include patients who had early discontinuation from the study.
  Change is calculated as End of Treatment (EOT) - Baseline
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set(FAS): all randomized patients who took at least 1 dose of double-blind study medication and had an assessment in OAB-q at both baseline and at least 1 post-baseline visit.
Measure: Number; unit: Participants
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 362 | 368
Participants
  Improvement from Baseline to End of Treatment | 231 | 278
  No Improvement from Baseline to End of Treatment | 131 | 90
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Test type: Superiority or Other; p = 0.0006, ANCOVA

5. Secondary Outcome: Patient Perception of Treatment Benefit at the End of Treatment in the Global Assessment Score of the Benefit, Satisfaction, and Willingness (BSW) Questionnaire
Description: The BSW questionnaire is a validated instrument that can be used to assess patient satisfaction with antimuscarinic agents for OAB. It is designed to capture the patient's perception of the effect of treatment in terms of relative benefit, patient satisfaction, and patient intention or willingness to continue on therapy.
Time Frame: Baseline and 12 Weeks
Population: The number assessed included all participants who completed the BSW questionnaire at baseline visit (visit 2) and end of treatment (visit 5/early withdrawal).
  A few patients who completed the BSW Questionnaire did not adequately complete the " Benefits" Section and therefore are considered 'N/A' for that Section.
Measure: Number; unit: Participants
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 316 | 335
Participants
  Benefit from Treatment - No | 115 | 53
  Benefit from Treatment - Little | 90 | 80
  Benefit from Treatment - Much | 109 | 196
  Benifit from Treatment - N/A | 2 | 6
  Satisfied with Treatment - No | 129 | 66
  Satisfied with Treatment - Yes | 187 | 269
  Willingness to Continue - No | 128 | 71
  Willingness to Continue - Yes | 188 | 264

6. Secondary Outcome: Change From Baseline to Each Visit in the OAB-q HRQL Sub-domain Scores of Coping, Concern, Sleep and Social
Description: The OAB-q is used to assess how much a patient is bothered by OAB symptoms & the impact on the patient's HRQL. It is comprised of 33 items, with raw scores for each sub-domain being converted to a scale of 0 to 100.
  Higher score values are indicative of better HRQL, and a positive score in change from baseline indicates improvement.
  Change is calculated End of Treatment (EOT) for each sub-domain - Baseline.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: Population is full analysis set(FAS): all randomized patients who took at least 1 dose of double-blind study medication and had an assessment in OAB-q at both baseline and at least 1 post-baseline visit.
  Number of participants analyzed per arm represents FAS. The numbers of participants for each visit/sub domain are noted in the category titles.
Measure: Mean (Standard Deviation); unit: OAB-q HRQL Sub Domain Score
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
OAB-q HRQL Sub Domain Score
  Coping- Baseline (N= 374 ; 377) | 53.7 (25.78) | 52.2 (26.76)
  Coping- Change at Week 4 (N=371; 370) | 14.9 (21.55) | 22.2 (22.20)
  Coping- Change at Week 8 (N=342; 356) | 18.9 (21.97) | 27.0 (24.81)
  Coping- Change at Week 12 (N=318; 339) | 19.9 (22.56) | 28.8 (25.22)
  Concern- Baseline (N= 374 ; 377) | 52.0 (25.49) | 51.9 (26.06)
  Concern- Change at Week 4 (N=371; 370) | 15.8 (21.58) | 22.4 (23.37)
  Concern- Change at Week 8 (N=342; 356) | 19.8 (22.87) | 28.4 (25.64)
  Concern- Change at Week 12 (N=318; 339) | 20.9 (23.10) | 29.9 (26.32)
  Sleep- Baseline (N= 374 ; 377) | 51.3 (25.78) | 47.3 (27.55)
  Sleep- Change at Week 4 (N=371; 370) | 13.9 (22.91) | 19.3 (23.68)
  Sleep- Change at Week 8 (N=342; 356) | 18.7 (24.46) | 26.2 (24.94)
  Sleep- Change at Week 12 (N=318; 339) | 19.0 (24.65) | 27.5 (26.56)
  Social- Baseline (N= 374 ; 377) | 78.9 (23.13) | 78.7 (23.56)
  Social- Change at Week 4 (N=371; 370) | 7.8 (16.51) | 10.3 (18.66)
  Social- Change at Week 8 (N=340; 356) | 9.4 (16.49) | 13.1 (19.65)
  Social- Change at Week 12 (N=318; 339) | 10.0 (17.81) | 13.7 (21.38)

7. Secondary Outcome: Change From Baseline in Work Productivity Assessment Index (WPAI)
Description: The WPAI is a tool used to evaluate the effect of solifenacin succinate on a patient's overall satisfaction & quality of life, and included 6 questions regarding the effect that bladder condition had on ability to perform work-related functions & carry out daily activities over the past 4 weeks. The scores were converted to percentages for reporting.
  A negative score in Change from Baseline indicates improvement. End of Treatment results include patients who had early discontinuation from the study.
  Change from baseline is based on the ANCOVA model after adjusting baseline value & center.
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set (FAS): all randomized patients who took at least 1 dose of double-blind study drug & had an OAB-q assessment at both baseline & at least 1 post-baseline visit.
  The number of participants analyzed per arm represents FAS. The numbers of participants for each timepoint / parameter are noted in the category titles.
Measure: Mean (Standard Deviation); unit: Percentage of indicated parameter
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
Percentage of indicated parameter
  % work time missed- Baseline (N=175;175) | 1.4 (8.60) | 1.1 (3.54)
  % work time missed- EOT (N=161;157) | 0.8 (5.85) | 0.5 (2.04)
  % work time missed- Change at EOT (N=145;142) | 0.1 (4.26) | -0.5 (3.34)
  % impairment while working- Baseline(N=203;194) | 27.5 (25.93) | 27.6 (25.72)
  % impairment while working- EOT (N=193;197) | 18.4 (21.11) | 13.2 (18.19)
  % impairment working-Change at EOT(N=172;175) | -8.7 (23.03) | -14.6 (24.09)
  % overall work impairment- Baseline (N=174;175) | 28.5 (25.77) | 28.2 (25.29)
  % overall work impairment- EOT (N=161;157) | 20.8 (21.81) | 14.1 (18.67)
  %overall work impairment-Change at EOT(N=145;142) | -8.2 (22.59) | -12.9 (23.00)
  %activity impairment- Baseline (N=368;375) | 38.6 (28.36) | 37.3 (27.44)
  % activity impairment- EOT (N=357;362) | 23.4 (23.17) | 19.2 (22.32)
  % activity impairment- Change at EOT(N=351;360) | -14.7 (25.46) | -18.1 (26.26)

8. Secondary Outcome: Change From Baseline in the Medical Care Use Index (MCUI) Medical Resource Utilization in the Past 3 Months
Description: MCUI is a Patient Reported Outcome instrument utilized to further evaluate the effect of solifenacin succinate on patient's overall satisfaction and quality of life.The tool included questions concerning the effect of the patients bladder condition on access to medical care.
  A negative score in Change from Baseline indicates improvement.
  End of Treatment results include patients who had early discontinuation from the study.
  Change is calculated as End of Treatment (EOT) - Baseline
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set(FAS):all randomized patients who took at least 1 dose of double-blind study medication & had an assessment in OAB-q at both baseline & at least 1 post-baseline visit. The number of participants analyzed per arm represents FAS. The numbers of participants for each timepoint/ parameter are noted in the category titles.
Measure: Mean (Standard Deviation); unit: Number of categorical items
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
Number of categorical items
  physician office visits- Baseline (N=371; 375) | 0.5 (1.30) | 0.5 (1.22)
  physician office visits- EOT (N=362; 366) | 0.2 (0.62) | 0.2 (0.79)
  physician office visits- Change at EOT(359; 365) | -0.4 (1.29) | -0.3 (1.23)
  urinary tract infections-Baseline (N=371; 370) | 0.1 (0.37) | 0.1 (0.46)
  urinary tract infections- EOT (N=358; 362) | 0.1 (0.28) | 0.1 (0.50)
  urinary tract infections-Change at EOT (355; 356) | -0.1 (0.38) | 0.0 (0.57)
  skin rashes- Baseline (N=367; 368) | 1.5 (10.52) | 0.3 (1.87)
  skin rashes- EOT (N=354; 357) | 1.0 (7.70) | 0.2 (1.83)
  skin rashes- Change at EOT (N=347; 351) | 0.0 (8.17) | -0.1 (1.63)
  falls- Baseline (N=365; 364) | 0.2 (0.86) | 0.2 (0.83)
  falls- EOT (N=356; 358) | 0.1 (0.72) | 0.5 (5.87)
  falls- Change at EOT (N=347; 349) | -0.1 (0.69) | 0.2 (5.83)
  pad/diapers used/ week- Baseline (N=371; 375) | 10.0 (19.17) | 10.4 (20.68)
  pad/diapers used/ week- EOT (N=360; 364) | 9.8 (24.07) | 8.3 (40.58)
  pad/diapers used/ week- Change at EOT(N=357; 362) | -0.2 (26.60) | -2.1 (42.01)

9. Secondary Outcome: Change From Baseline in the MCUI Behavior Therapy Stratified
Description: MCUI is a Patient Reported Outcome instrument utilized to further evaluate the effect of solifenacin succinate on patient's overall satisfaction and quality of life. The tool included questions concerning the effect of the patients bladder condition on access to medical care.
  A negative score in Change from Baseline indicates improvement.
  End of Treatment results include patients who had early discontinuation from the study.
  Change is calculated as End of Treatment (EOT) - Baseline
Time Frame: Baseline and 12 Weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
Number of Days
  days with timed voiding- Baseline (N=364; 365) | 14.8 (37.33) | 12.1 (29.35)
  days with timed voiding- EOT (N=356; 360) | 10.3 (27.07) | 7.4 (23.13)
  days with timed voiding-Change at EOT(N=347; 350) | -4.0 (37.38) | -5.3 (33.66)
  days with fluid management-Baseline(N=368; 369) | 21.3 (40.07) | 22.1 (38.38)
  days with fluid management- EOT (N=355; 366) | 15.1 (28.76) | 11.5 (25.10)
  days with fluid management-Change at EOT(349; 360) | -6.3 (42.36) | -11.0 (40.43)
  days w/ pelvic floor exercises-Baseline(364; 366) | 8.5 (22.17) | 9.2 (22.78)
  days w/ pelvic floor exercises- EOT (N=352; 358) | 12.1 (56.94) | 5.5 (17.31)
  days w/pelvic flr exercises-Change atEOT(344; 349) | 3.4 (50.96) | -3.2 (19.43)
  days with biofeedback- Baseline (N=359; 360) | 0.4 (5.32) | 0.1 (0.95)
  days with biofeedback- EOT (N=352; 358) | 0.0 (0.53) | 0.0 (0.45)
  days with biofeedback- Change at EOT (N=338; 343) | -0.4 (5.18) | 0.0 (1.08)
  days w/ electrical stimulation-Baseline (358; 362) | 0.0 (0.63) | 0.1 (1.58)
  days w/ electrical stimulation- EOT (N=352; 358) | 0.0 (0.43) | 0.1 (0.56)
  days w/ elec stimulation-Change at EOT(N=337; 345) | 0.0 (0.79) | 0.0 (1.68)

10. Secondary Outcome: Change From Baseline in International Consultation on Incontinence Modular Questionnaire Male Sexual Matters Associated With Lower Urinary Tract Symptoms (ICIQ-MLUTSsex) Overall Symptom and Bother Scores.
Description: ICIQ-MLUTSsex is a patient reported outcome instrument to further evaluate the effect of solifenacin succinate on patients' overall satisfaction & quality of life. The questionnaire contains 5 questions for detailed evaluation of sexual matters associated with lower urinary track symptoms & impact on sexual quality of life, with a scale of 0 to 12.
  Change from baseline with a negative score indicates improvement. End of Treatment results include patients who had early discontinuation. Change is calculated as End of Treatment(EOT)-Baseline.
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set(FAS): all randomized male patients who took at least 1 dose of double-blind study medication and had an assessment in OAB-q at both baseline and at least 1 post-baseline visit.
  The number of participants analyzed per arm represents FAS. The numbers of participants for each visit are noted in the category titles.
Measure: Mean (Standard Deviation); unit: ICIQ-MLUTSsex
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 60 | 71
ICIQ-MLUTSsex
  Symptom- Baseline (N=59; 71) | 3.6 (2.81) | 3.5 (3.01)
  Symptom- EOT (N=55; 68) | 3.2 (2.71) | 3.7 (3.00)
  Symptom- Change at EOT (N=54; 68) | -0.1 (1.57) | 0.1 (1.87)
  Bother- Baseline (N=59; 71) | 12.1 (11.47) | 11.8 (11.21)
  Bother- EOT (N=51; 67) | 10.3 (10.53) | 11.4 (11.17)
  Bother- Change at EOT (N=50; 67) | -1.6 (8.24) | -0.6 (9.32)

11. Secondary Outcome: Change From Baseline in International Consultation on Incontinence Modular Questionnaire Female Sexual Matters Associated With Lower Urinary Tract Symptoms (ICIQ-FLUTSsex)Overall Symptom and Bother Scores.
Description: ICIQ-FLUTSsex is a patient reported outcome instrument to further evaluate the effect of solifenacin succinate on patients' overall satisfaction & quality of life.The questionnaire contains 5 questions for detailed evaluation of sexual matters associated with lower urinary track symptoms & impact on sexual quality of life, with a scale of 0 to 14.
  Change from baseline with a negative score indicates improvement. End of Treatment results include patients who had early discontinuation. Change is calculated as End of Treatment(EOT)-Baseline.
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set(FAS): all randomized female patients who took at least 1 dose of double-blind study medication and had an assessment in OAB-q at both baseline and at least 1 post-baseline visit.
  The number of participants analyzed per arm represents FAS. The numbers of participants for each visit are noted in the category titles.
Measure: Mean (Standard Deviation); unit: ICIQ-FLUTSsex
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 314 | 306
ICIQ-FLUTSsex
  Symptom- Baseline (N=302; 300) | 4.9 (3.69) | 5.2 (3.63)
  Symptom- EOT (N=297; 291) | 3.9 (3.46) | 3.8 (3.55)
  Symptom- Change at EOT (N=288; 288) | -0.9 (3.53) | -1.3 (3.75)
  Bother- Baseline (N=281; 282) | 9.0 (10.77) | 10.0 (11.47)
  Bother- EOT (N=263; 262) | 6.1 (8.52) | 6.6 (9.43)
  Bother- Change at EOT (N=245; 249) | -3.1 (8.11) | -3.6 (9.04)

12. Secondary Outcome: Change From Baseline in the Treatment Satisfaction Visual Analog Scale (TS-VAS)
Description: The TS-VAS is a instrument utilized to further evaluate the effect of solifenacin succinate on patients' overall satisfaction & quality of life. Each patient completed a TS-VAS to rate satisfaction with treatment. They were to answer the following question: "Are you satisfied with your treatment?" by placing a mark on a line that ran from 0 (no, not at all) to 100 (yes, completely).
  Change from baseline with a positive score indicates an improvement. The End of Treatment (EOT) results include patients who had early discontinuation from the study.
  Change is calculated as EOT - Baseline
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set(FAS): all randomized patients who took at least 1 dose of double-blind study medication and had an assessment in OAB-q at both baseline and at least 1 post-baseline visit.
  The number of participants analyzed per arm represents FAS. The numbers of participants for each row are noted in the category titles.
Measure: Mean (Standard Deviation); unit: TS-VAS
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
TS-VAS
  Baseline (N=363; 367) | 32.7 (35.29) | 29.0 (33.99)
  End of Treatment (N=363; 367) | 51.2 (38.10) | 67.4 (34.38)
  Change at EOT (N=352; 357) | 18.4 (47.28) | 38.2 (45.38)
Statistical Analysis 1: Comparison: Placebo vs Solifenacin Succinate; Statistical Analysis applies to 'Change at EOT'; Test type: Superiority or Other; p < .0001, ANCOVA; Least Square Mean Difference = -16.8, 95% CI [-22.1 to -11.6]

13. Secondary Outcome: Change From Baseline to End of Treatment in Mean Parameters Per 24 Hours Recorded in 3-day Diary
Description: The mean parameters recorded for previous 24 hours in the 3-day diary were: number of micturitions, number of incontinence episodes, number of urgency episodes, number of nocturia episodes and number of nocturnal voids.
  Change from baseline with a lower score indicates an improvement.
  End of Treatment (EOT) results include patients who had early discontinuation from the study; only patients who had the symptom at baseline and data at the EOT in the 3-day diary are included in the data table.
  Change is calculated as EOT - Baseline
Time Frame: Baseline and 12 Weeks
Population: Population is full analysis set(FAS): all randomized patients who took at least 1 dose of double-blind study drug & had an OAB-q assessment at both baseline & at least 1 post-baseline visit.
  The number of participants analyzed per arm represents FAS. The number of participants for each timepoint / parameter are noted in the category titles.
Measure: Mean (Standard Deviation); unit: Number of Category Events / 24 Hours
Arm/Group | Placebo | Solifenacin Succinate
Number analyzed (Participants) | 374 | 377
Number of Category Events / 24 Hours
  Micturitions- Baseline (N=363;369) | 11.85 (4.039) | 11.73 (3.693)
  Micturitions- End of Treatment (N=363;369) | 10.49 (3.645) | 9.50 (3.869)
  Micturitions- Change at EOT (N=363;369) | -1.36 (3.203) | -2.23 (3.482)
  Incontinence Episodes- Baseline (N=267;268) | 2.80 (2.584) | 2.92 (2.743)
  Incontinence Episodes-End of Treatment (N=267;268) | 1.56 (2.338) | 1.07 (2.156)
  Incontinence Episodes-Change at EOT (N=267;268) | -1.24 (2.545) | -1.85 (2.484)
  Urgency Episodes- Baseline (N=364;369) | 5.70 (3.895) | 5.72 (3.734)
  Urgency Episodes- End of Treatment (N=364;369) | 3.86 (3.795) | 2.66 (3.381)
  Urgency Episodes- Change at EOT (N=364;369) | -1.84 (3.891) | -3.05 (3.932)
  Nocturia Episodes- Baseline (N=309;313) | 1.57 (0.968) | 1.74 (1.191)
  Nocturia Episodes- End of Treatment (N=309;313) | 1.09 (1.025) | 1.11 (1.241)
  Nocturia Episodes- Change at EOT (N=309;313) | -0.48 (1.015) | -0.63 (1.132)
  Nocturnal Voids- Baseline (N=329;326) | 1.89 (1.429) | 1.99 (1.520)
  Nocturnal Voids- End of Treatment (N=329;326) | 1.41 (1.299) | 1.29 (1.352)
  Nocturnal Voids- Change at EOT (N=329;326) | -0.48 (1.542) | -0.70 (1.513)

ADVERSE EVENTS:
Arm/Group | Placebo | Solifenacin Succinate
Serious Adverse Events (participants affected / at risk) | 6/382 | 3/386
Other Adverse Events (participants affected / at risk) | 18/382 | 84/386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=382) | Solifenacin Succinate (N=386)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Migration of Implant (General disorders) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Ammonia Increased (Investigations) | 1 | 0
Hypokalaemia (Investigations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Discitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ruptured Cerebral Aneurysm (Nervous system disorders) | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=382) | Solifenacin Succinate (N=386)
Constipation (Gastrointestinal disorders) | 9 | 32
Dry Mouth (Gastrointestinal disorders) | 9 | 52

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.